CLINICAL TRIAL: NCT03807622
Title: A Prospective, Nonrandomized, Non-interventional Trial to Evaluate ClearSight System Cardiac Output in China
Brief Title: ClearSight System CHN Study
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-05
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Patient With Clinically Indicated Invasive Monitoring
Keywords: Elective Major Cardiothoracic; Mitral Valve Surgery; Coronary Artery Bypass Grafting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: EV1000NI Clinical Platform: Noninvasive Hemodynamic Monitoring utilizing ClearSight System — EV1000NI Clinical Platform: Noninvasive Hemodynamic Monitoring utilizing ClearSight System

SUMMARY:
The purpose of this clinical trial is to demonstrate that cardiac output (CO) as determined with the Clinical Platform (Model:EV1000A, Software Version:1.9) in a noninvasive manner is comparable to CO as determined by Pulmonary Artery Catheter (PAC) thermodilution (TD). The results of this study may be used for registration and regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age
* Subjects provide written informed consent prior to trial procedures
* Subjects' height and weight must be accurately obtained prior to study start.

Exclusion Criteria:

* Aortic or tricuspid valve regurgitation
* Aortic stenosis or aneurysms
* Cardiac rhythm disorder
* Patients with extreme contraction of the smooth muscle in the arteries and arterioles in the lower arm and hand, such as may be present in patients with Raynaud's or Buerger's disease or with extremely cold hands
* Inability to place the finger cuff appropriately due to subject anatomy or condition
* Known pregnancy
* Patients being treated with an intra-aortic balloon pump
* Patient is currently participating in an investigational drug or another device study that clinically interferes with the study endpoints
* Intracardiac shunt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major cardiothoracic surgery with an indwelling PA catheter. The surgical intervention includes, but is not limited to, mitral valve surgery or coronary artery bypass grafting.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-12-25 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Cardiac Output using the Non-invasive ClearSight System | Expected to last no more than 6 hours
  Cardiac Output using the Non-invasive ClearSight System

SECONDARY OUTCOMES:
The percentage error (PE) between the ClearSight System CO and TD | Expected to last no more than 6 hours
  The percentage error (PE) between the ClearSight System CO and TD

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Fuwai Cardiovascular Disease Hospital, Chinese Academy of Medical Sciences, Beijing, Xicheng, Beijing Municipality
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Tianjin Chest Hospital, Xiaobailou, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Y, Huang W, Han J, Tian Y, Wang C, Li L. A comparison of ClearSight noninvasive cardiac output and pulmonary artery bolus thermodilution cardiac output in cardiac surgery patients. Perioper Med (Lond). 2022 Jun 9;11(1):24. doi: 10.1186/s13741-022-00248-1. PMID 35676705